CLINICAL TRIAL: NCT03253003
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2017_27
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Sonova2017_27
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Hearing Loss, Bilateral Sensorineural, Progressive
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: A line extension of the Phonak Audéo B hearing aid product family will be fitted to the participants individual hearing loss.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Audéo B hearing aid line extension (Experimental): The line extension of the Phonak Audéo B product family will be fitted to the participants individual hearing loss.
  Interventions: Device: Line extension of the Phonak Audéo B product family

INTERVENTIONS:
Device: Line extension of the Phonak Audéo B product family — The line extension of Phonak Audéo B product family will be fitted to the participants individual hearing loss.

SUMMARY:
A methodical evaluation of new CE-labelled Phonak Hearing Systems is intended to be conducted on hard of participants with a hearing loss to grant quality control prior to product launch. The aim of the investigation series is to ensure a stable overall performance of the new hearing systems, a good sound quality during phone calls as well as maximum benefit for the participant with the devices.

DETAILED DESCRIPTION:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials in the way as planned for this study ("phase of final inspection"). This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years) with and without (experience with) hearing aids
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Informed Consent as documented by signature
* Smartphone user

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Central hearing disorders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Stable performance in daily life | Three weeks
  The data, serving as primary outcomes are collected in a series of home trials, taking place between the lab trial appointments. The stable performance in daily life (that means: no significant interruptions, distortions, artefacts, feedback, system noise or other malfunctions) will be assessed with the aid of quantitative questionnaires. Descriptive statistics will be executed. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.
Phone call - Sound Quality | One week
  The data serving as primary outcomes are collected in a lab appointment. The participants will be asked to have a phone call with the investigator in the lab. The sound quality will be subjectively assessed by the participants and additionally by the investigators on given scales. Descriptive statistics will be executed. Interference statistics will be executed by applying the appropriate parametric or non-parametric test, depending on the data's distribution. A significance level of 5% is pursued.

CONTACTS AND LOCATIONS:
Overall Officials: Simone Ebbing, B. Sc., Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No